CLINICAL TRIAL: NCT04970719
Title: The Efficacy of Baricitinib Plus Remdesivir Compared to Dexamethasone Plus Remdesivir in Hospitalised COVID-19 Patients With Diabetes Mellitus
Brief Title: Baricitinib in Hospitalized Covid-19 Patients With Diabetes Mellitus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: adequate cases were not available
Sponsor: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other)
Responsible Party: Principal Investigator, Wasim Md Mohosin Ul Haque, Associate Professor, Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BADAS-ERC/EC/21/00311
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; baricitinib; remdesivir; dexamethasone; diabetes mellitus; hospitalized
MeSH Terms: conditions — COVID-19; Diabetes Mellitus | interventions — baricitinib; Janus Kinase Inhibitors; Dexamethasone; Steroids; remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remdesivir plus Baricitinib (Experimental): 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 5-day total course; 4 mg of baricitinib administered as 2 tablets taken orally daily while hospitalized for up to a 14-day total course
  Interventions: Drug: Baricitinib; Drug: Remdesivir
- Remdesivir plus Dexamethasone (Active Comparator): 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 5 -day total course; and 6 mg of dexamethasone administered as an intravenous injection daily while hospitalized for up to a 10-day total course.
  Interventions: Drug: Dexamethasone; Drug: Remdesivir

INTERVENTIONS:
Drug: Baricitinib — 4 mg of baricitinib administered as 2 tablets taken orally daily while hospitalized for up to a 14-day total course
  Other Names: Janus kinase inhibitors
  Arms: Remdesivir plus Baricitinib
Drug: Dexamethasone — and 6 mg* of dexamethasone administered as an intravenous injection daily while hospitalized for up to a 10-day total course
  Other Names: Steroids
  Arms: Remdesivir plus Dexamethasone
Drug: Remdesivir — 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of remdesivir while hospitalized for up to a 5-day total course
  Other Names: Anti-viral

SUMMARY:
To date, some of the most promising drugs used in the treatment of COVID pneumonia are systemic corticosteroids, remdesivir and baricitinib. Dexamethasone has been found efficacious in reducing mortality in patients requiring supplemental oxygen and mechanical ventilation. There is a trend towards reduced mortality in patients who receive remdesivir and dexamethasone combination, supporting the hypothesis that an antiviral drug combined with an anti-inflammatory agent improve outcomes in COVID-19. Baricitinib plus remdesivir is superior to remdesivir alone in reducing recovery time and accelerating improvement in clinical status among patients with COVID-19, notably among those receiving high-flow oxygen non-invasive ventilation. Diabetes mellitus increases the risk for COVID-19 morbidity and mortality. Patients with diabetes have coexisting morbidities and already immune-compromised. Steroids cause further immunosuppression and may contribute to uncontrolled blood glucose in this group of patients, resulting in worse outcomes. Baricitinib can be an alternative to corticosteroids in diabetic patients. This open-label multi-centre non-inferiority randomized controlled trial will be conducted in seven hospitals in Bangladesh. The primary objective is to evaluate the clinical efficacy of baricitinib plus remdesivir compared to dexamethasone plus remdesivir in hospitalized COVID-19 patients with diabetes mellitus, as assessed by the proportion of patients, need "rescue treatment" between two groups by day 29. Hospitalized adult (≥18 years) diabetic patients with confirmed SARS-CoV-2 infection have ordinal scale category 5 will be included in the study. Subjects will be randomized in a 1:1 (by tossing a coin) ratio in two groups. The total sample size is 362. Group 1 subjects will receive 200 mg of remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily dose of remdesivir while hospitalized for up to 5 days and 4 mg of baricitinib administered as 2 tablets taken orally daily while hospitalized for up to 14 days. Group 2 will receive the same dose of remdesivir plus 6 mg of dexamethasone administered as an intravenous injection daily while hospitalized for up to 10 days. Subjects will be assessed daily while hospitalized. Discharged subjects will be evaluated on days 15, 22 and 29 (in person; if not possible, over the telephone). Assessment will be done clinically using an 8-point Ordinal Scale and National Early Warning Score.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which was first identified during an outbreak of a respiratory illness in Wuhan City of Hubei Province, China, in December 2019. On March 11, WHO declared COVID-19 a global pandemic. COVID-19 situation is sprouting rapidly with increasing case counts and deaths. So far (June 29, 2021), 182.2 million cases have been detected, with 3.95 million deaths worldwide. . High infection and case fatality rates warrant ongoing research to find safe and effective treatment protocols for hospitalized patients. To date, some of the most promising drugs used in treating COVID pneumonia are systemic corticosteroids, remdesivir and baricitinib. The first randomized clinical trial of remdesivir did not show an absolute decrease in mortality. Subsequently, the ATCC-1 trial conclusively demonstrated a benefit. A third open-label trial involvingCOVID-19 with moderate severity had a low overall mortality (<2%) and did not provide further insight. Finally, data from the SOLIDARITY trial, the largest remdesivir trial to date with 5451 patients (WHO Solidarity Trial Consortium, 2021), did not show a significant decrease in mortality for remdesivir alone (rate ratio 0.95, 95% CI 0.81-1.11) or their embedded meta-analysis of all available trials (rate ratio 0.91, 95% CI 0.79-1.05).Though remdesivir showed promising clinical benefit, the high mortality in the ATCC-1 trial underscored using an immunomodulator combined with remdesivir to achieve the desired outcome . There was a trend towards reduced mortality in patients who received remdesivir and dexamethasone combination. This observation supports the hypothesis that the combination of antiviral and anti-inflammatory agents could improve the outcomes of COVID-19.

Baricitinib is an inhibitor of Janus kinase (JAKs) 1 and 3, with partial selectivity to JAK 2. Baricitinib suppresses pro-inflammatory signals that may be pathogenetically important in the progression to more severe lung disease and ARDS in patients with COVID-19. So far, dexamethasone and baricitinib are the only two anti-inflammatory treatment options; those have been shown to be effective in large randomized clinical trials in treating adults with COVID-19 in hospitals. However, differences in study populations, mortality rates, and endpoint data collected in the ACTT-2 and RECOVERY studies make it difficult to draw firm conclusions about the value of interventions in different patient populations. A comparison between baricitinib and dexamethasone for treating patients with COVID-19 pneumonia who require supplemental oxygen is now a fascinating topic for clinical research, mentioned in an editorial in the New England Journal of Medicine.

ACTT-2showed that baricitinib plus remdesivir was superior to remdesivir alone in reducing recovery time and accelerating improvement in clinical status among patients with COVID-19, notably among those receiving high-flow oxygen or non-invasive ventilation. The combination was associated with fewer serious adverse events like serious infections.Baricitinib was most effective in patients with an ordinal scale of 5 and 6, allowing expansion of therapeutic armament against COVID-19 pneumonia, mainly in patients receiving oxygen support without invasive mechanical ventilation.Evidence in favour of baricitinib is emerging; a recent meta-analysis and systematic review of five studies with a total of 1190 patients showed that the use of JAK inhibitors was significantly associated with a reduced risk of mortality (OR=0.51; 95% CI, 0.28 to 0.93; P = 0.02; I2: 7.8%, P = 0.354) and clinical improvement (OR=1.76; 95% CI, 1.05 to 2.95; P = 0.032; I2: 26.4%, P = 0.253) . Another systematic review of 6 cohort studies and 5 clinical trials involving 2367 subjects treated with ruxolitinib (N = 3) or baricitinib (N = 8) found a potential role for JAK-inhibitors in reducing the risk of death in persons with COVID-19. Use of JAK-inhibitors decreased use of invasive mechanical ventilation (RR = 0.63; 95% CI, 0.47 to 0.84; P = 0.002) and had borderline impact on rates of ICU admission (RR = 0.24; 95% CI, 0.06 to 0.02; P = 0.05) and ARDS (RR = 0.50; 95% CI, 0.19 to1.33; P = 0.16). Relative risks of death for both drugs were 0.42; 95% CI, 0.30 to 0.59; P < 0.001, for ruxolitinib, RR = 0.33; 95% CI, 0.13 to 0.88; P = 0.03) and for baricitinib RR = 0.44; 95% CI, 0.31 to 0.63; P < 0.001). A recent Brazilian study found that tofacitinib resulted in a lower risk of death or respiratory failure than placebo in patients hospitalized with Covid-19 pneumonia.

Dexamethasone has been established as life-saving by reducing mortality in patients needing supplemental oxygen and mechanical ventilation . Dexamethasone was evaluated at the University of Oxford-sponsored Global Study on the Randomised Evaluation of COVID-19 Therapy (RECOVERY). The study results showed that patients receiving dexamethasone had a lower death rate than patients receiving usual treatment. However, in this study, no ordinal stratification was used. The mortality benefit of dexamethasone was greater in patients receiving invasive mechanical ventilation. (assumed ordinal scale of 7). Nevertheless, no indication of the level of oxygen support was given; therefore, it is unknown whether dexamethasone was effective in patients who received low flow oxygen (ordinal scale 5) or in patients who received high flow oxygen (ordinal scale 6).

To date, ACTT-4 is the only head to head study comparing these two drugs in a similar population. The preliminary report of this study is equivocal. No differences in efficacy or adverse reactions were found between the two groups; no drugs were found to be superior or inferior to one another.

Dexamethasone is associated with high blood glucose levels, especially in patients with diabetes, and often gets out of hand. Recent retrospective analyses of hospitalized patients have strongly suggested that "diabetes" increases the risk for COVID-19 morbidity and mortality. Another study found that patients with COVID-19 who have elevated blood glucose levels without a previous diagnosis of diabetes may be at a high risk of death and an increased risk of severe complications. The recent surge of mucormycosis in diabetic COVID-19 is supposed to be a consequence of using high dose steroids in this patient population.

Diabetic patients often have other concomitant comorbidities and are already immunosuppressed. High dose steroids lead to additional immunosuppression with uncontrolled blood glucose in this group of patients, leading to a worse outcome. Baricitinib may be a reasonable alternative to dexamethasone in diabetic patients. This drug has already been recommended for COVID-19 patients with grossly uncontrolled diabetes. The present study aims to compare the outcome between patients treated with dexamethasone plus remdesivir and baricitinib plus remdesivir in the diabetic population. This study will help clinicians contextualize the evidence and practice sane medicine when selecting drugs to treat COVID-19 patients with coexisting diabetes mellitus.

Research question:

Is baricitinib plus remdesivir as effective as dexamethasone plus remdesivir in hospitalized diabetic patients with COVID-19?

Hypothesis:

Baricitinib plus remdesivir is not less effective than dexamethasone plus remdesivir in hospitalized diabetic patients with COVID-19.

Study design:

Open-label, multi-centre randomized controlled non-inferiority trial. Randomization: 1:1 (by tossing a coin). Non-Inferiority margin: M1=1.0309, M2=1.0153.

Assessment procedure:

* Subjects will be assessed daily while hospitalized.
* For discharged subjects Day 15 and 29 (in person; if not possible, over the telephone) Physical and biochemical examination The Day 22 (over the telephone) Only clinical data
* Al patient-related data will be updated in a web-based structured form instantly

Assessment tools

* Clinical

  1. 8-point Ordinal scale activities and no new or increased oxygen use.
  2. National Early Warning Score 2 (NEWS 2, table 2)
* Laboratory:

CBC, HbA1c, fasting blood glucose, CRP, serum ferritin, LDH, D-dimer, serum creatinine, SGPT, SGOT, PT/APTT, serum procalcitonin, serum electrolytes, serum fibrinogen, IL-6 level, blood and sputum culture and sensitivity, imaging.

Assessment frequency

* Clinical: daily during hospitalization, after discharge on day 15, 22, and 29.
* Biochemical:

  * CRP: 24 hourly for 1st48 hours of randomization, then on day 3, 5, 8, 11, 15, and 29.
  * CBC, serum ferritin, LDH, D-dimer, serum creatinine, SGPT, SGOT, fasting blood glucose on randomization and day 3, 5, 8, 11, 15, and 29.
  * HbA1c, PT/APTT, serum procalcitonin, total serum bilirubin, on the day of randomization then as relevant.
  * Serum fibrinogen level, serum IL-6 level, serum electrolytes relevant.
* Microbiological tests:

  o Blood and sputum culture and sensitivity as relevant
* Imaging:

  * CXR on the day of randomization and as relevant.
  * HRCT as relevant.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized diabetic adults with laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) in any respiratory specimen within 10 days prior to randomization or *Hospitalized diabetic adults with typical features of COVID-19 for 10 days prior to randomization, not yet tested for SARS-CoV-2 infection by PCR in any respiratory specimen.

  * RT-PCR for SARS-CoV-2 will be performed within 48 hours of enrollment and excluded from the study if found to be negative.
* 8-point ordinal scale "category 5" patients, but O2 requirement not more than 10L / min.
* The subject provides informed consent before initiating any study procedures and understands and agrees to comply with planned study procedures

Exclusion Criteria:

* Patients with evidence (clinical, hematological, microbiological or imaging ) of sepsis or any acute/subacute coinfection at the time of enrollment.
* Patients who have already received any of the study drugs prior to randomization.
* Patients with severe renal and/or hepatic impairment (eGFR <30 mL/min [EPI-CKD formula] or serum ALT more than 5 times normal upper limit, serum bilirubin > 2 mg/dl).
* Patients with known COPD.
* Patients with absolute neutrophil count <700 cells/microliter, 0.7 x 103/microliter.
* Patients with absolute lymphocyte count <200 cells/microliter, 0.20 x 103/microliter.
* Patients who are allergic to any of the study drugs.
* Patients with chronic infections, such as tuberculosis (TB), HIV infection etc.
* Immunosuppressed patients, such as taking cytotoxic/immunomodulating drugs or systemic steroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rescue treatment | Day 2 through Day 29
  The proportion of subjects not requiring "rescue treatment".
  Rescue treatment will be given if there is a deterioration of the ordinal scale beyond category 5 (unable to maintain SpO2 ≥ 92% with 10 L/ min O2) at any time 24 hours after enrollment.
  10 mg of dexamethasone will be administered on top of existing treatment in group 1 and escalate to in group 2 as an intravenous injection, 2 to 4 times daily for 3 to 5 days based on the patient's condition, then tapered.
  Patients who deteriorate beyond the ordinal scale category 5 within 24 hours of enrollment will be excluded from the study.

SECONDARY OUTCOMES:
Death or invasive mechanical ventilation | Day 2 through Day 29
  The proportion of subjects not meeting criteria for one of the following two ordinal scale categories at any time: 8) Death; 7) Hospitalized, on invasive mechanical ventilation
C-reactive protein (CRP) | Day 1 through Day 29
  Change from baseline in C-reactive protein (CRP)
lactate dehydrogenase (LDH) | Day 1 through Day 29
  Change from baseline in lactate dehydrogenase (LDH)
Ferritin | Day 1 through Day 29
  Change from baseline in Ferritin
Creatinine | Day 1 through Day 29
  Change from baseline in creatinine
alanine aminotransferase (ALT) | Day 1 through Day 29
  Change from baseline in alanine aminotransferase (ALT)
d-dimer concentration | Day 1 through Day 29
  Change from baseline in d-dimer concentration
fasting blood glucose (FBS) | Day 1 through Day 29
  Change from baseline in fasting blood glucose (FBS)
hemoglobin | Day 1 through Day 29
  Change from baseline in hemoglobin
platelets | Day 1 through Day 29
  Change from baseline in platelets
white blood cell count (WBC) | Day 1 through Day 29
  Change from baseline in white blood cell count (WBC)
total lymphocyte count | Day 1 through Day 29
  Change from baseline in total lymphocyte count
adverse events (AEs) | Day 1 through Day 29
  Cumulative incidence of Grade 3 and 4 clinical and/or laboratory adverse events (AEs)
serious adverse events (SAEs) | Day 1 through Day 29
  Cumulative incidence of serious adverse events (SAEs) An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect Grade 3 AEs are defined as events that interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as events that are potentially life threatening.
invasive mechanical ventilation | Day 2 through Day 29
  Days of invasive mechanical ventilation (if applicable)
non-invasive ventilation/high flow oxygen | Day 2 through Day 29
  Days of non-invasive ventilation/high flow oxygen (if applicable)
supplemental oxygen | Day 1 through Day 29
  Days of supplemental oxygen
Desirability of Outcome Ranking (DOOR) | Day 15 through Day 29
  Desirability of Outcome Ranking (DOOR) based on ordinal scale: 1) Recovered (category 1, 2 or 3 on ordinal scale); 2) Improved (> / = 1 category improvement of ordinal scale compared with baseline) & no serious adverse event (SAE); 3) Improved (> / = 1 category improvement of the ordinal scale compared with baseline) & SAE (related or unrelated); 4) No change in ordinal scale from baseline & no SAE; 5) No change in ordinal scale from baseline & SAE (related or unrelated); 6) Worsening (> / = 1 category worse in ordinal scale from baseline); 7) Death.
Duration of hospitalization | Day 1 through Day 29
  Measured in days
Incidence of discontinuation or temporary suspension of study product administration | Day 1 through Day 10
  For any reason
Subject 14-day mortality | Day 2 through Day 15
  Date of death (if applicable).
Subject 28-day mortality | Day 2 through Day 29
  Date of death (if applicable).
Subject clinical status | Days 3, 5, 8, 11, 15, 22, and 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use
The proportion of subjects meeting criteria for each of the 8 ordinal scale categories | Day 15
  The ordinal scale categories are defined as: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use
The proportion of subjects not meeting criteria for one of the three most severe ordinal scale categories at any time | Day 2 through Day 29
  The ordinal scale categories: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices.
Time to an improvement of one category from baseline using an ordinal scale | Day 1 through Day 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, but has a new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, the patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use.
Time to recovery | Day 1 through Day 29
  Day of recovery is defined as the first day on which the subject satisfies one of the following three ordinal scale categories: 3) Hospitalized, not requiring supplemental oxygen and no longer requires ongoing medical care; 2) Not hospitalized, but has new or increased limitation on activities and/or new or increased requirement for home oxygen over baseline, pre-COVID-19 status; 1) Not hospitalized, patient is back to their baseline, pre-COVID-19 status, that is, no new or increased limitations on activities and no new or increased oxygen use.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim MM Haque, FCPS, Principal Investigator — Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders
Locations (7):
- Bangladesh (7):
  - Debidwar Upazila Health Complex, Comilla
  - BIRDEM General Hospital, Dhaka
  - Mugda Medical College and Hospital, Dhaka
  - Kurmitola General Hospital, Dhaka
  - Kurigram Adhunik Sadar Hospital, Kurigrām
  - Rajshahi Medical College & Hospital, Rajshahi
  - Dedicated Corona Isolation Hospital (DCIH), Rangpur City

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: relative to the time when summary data are published
Access Criteria: all data will be available if required

REFERENCES:
- [Background] Ahmed SB, Dumanski SM. Sex, gender and COVID-19: a call to action. Can J Public Health. 2020 Dec;111(6):980-983. doi: 10.17269/s41997-020-00417-z. Epub 2020 Sep 29. PMID 32990927
- [Background] Cucinotta D, Vanelli M. WHO Declares COVID-19 a Pandemic. Acta Biomed. 2020 Mar 19;91(1):157-160. doi: 10.23750/abm.v91i1.9397. PMID 32191675
- [Background] Goletti D, Cantini F. Baricitinib Therapy in Covid-19 Pneumonia - An Unmet Need Fulfilled. N Engl J Med. 2021 Mar 4;384(9):867-869. doi: 10.1056/NEJMe2034982. No abstract available. PMID 33657299
- [Background] NIH closes enrollment in trial comparing COVID-19 treatment regimens: National Institutes of Health 2021 [updated April 15. Available from: https://www.nih.gov/news-events/news-releases/nih-closes-enrollment-trial-comparing-covid-19-treatment-regimens.
- [Background] Natanegara F, Zariffa N, Buenconsejo J, Ran L, Cooner F, Lakshminarayanan D, et al. Statistical Opportunities to Accelerate Development for COVID-19 Therapeutics. Statistics in Biopharmaceutical Research. 2020:1-17.
- [Background] Smith GB, Redfern OC, Pimentel MA, Gerry S, Collins GS, Malycha J, Prytherch D, Schmidt PE, Watkinson PJ. The National Early Warning Score 2 (NEWS2). Clin Med (Lond). 2019 May;19(3):260. doi: 10.7861/clinmedicine.19-3-260. No abstract available. PMID 31092526
- [Background] Coronavirus Disease 2019 (COVID-19) Treatment Guidelines [Internet]. Bethesda (MD): National Institutes of Health (US); 2021 Apr 21-2024 Mar 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK570371/ PMID 34003615
- [Result] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Result] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Result] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Result] Kalil AC, Patterson TF, Mehta AK, Tomashek KM, Wolfe CR, Ghazaryan V, Marconi VC, Ruiz-Palacios GM, Hsieh L, Kline S, Tapson V, Iovine NM, Jain MK, Sweeney DA, El Sahly HM, Branche AR, Regalado Pineda J, Lye DC, Sandkovsky U, Luetkemeyer AF, Cohen SH, Finberg RW, Jackson PEH, Taiwo B, Paules CI, Arguinchona H, Erdmann N, Ahuja N, Frank M, Oh MD, Kim ES, Tan SY, Mularski RA, Nielsen H, Ponce PO, Taylor BS, Larson L, Rouphael NG, Saklawi Y, Cantos VD, Ko ER, Engemann JJ, Amin AN, Watanabe M, Billings J, Elie MC, Davey RT, Burgess TH, Ferreira J, Green M, Makowski M, Cardoso A, de Bono S, Bonnett T, Proschan M, Deye GA, Dempsey W, Nayak SU, Dodd LE, Beigel JH; ACTT-2 Study Group Members. Baricitinib plus Remdesivir for Hospitalized Adults with Covid-19. N Engl J Med. 2021 Mar 4;384(9):795-807. doi: 10.1056/NEJMoa2031994. Epub 2020 Dec 11. PMID 33306283
- [Result] Wang Y, Zhang D, Du G, Du R, Zhao J, Jin Y, Fu S, Gao L, Cheng Z, Lu Q, Hu Y, Luo G, Wang K, Lu Y, Li H, Wang S, Ruan S, Yang C, Mei C, Wang Y, Ding D, Wu F, Tang X, Ye X, Ye Y, Liu B, Yang J, Yin W, Wang A, Fan G, Zhou F, Liu Z, Gu X, Xu J, Shang L, Zhang Y, Cao L, Guo T, Wan Y, Qin H, Jiang Y, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Remdesivir in adults with severe COVID-19: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2020 May 16;395(10236):1569-1578. doi: 10.1016/S0140-6736(20)31022-9. Epub 2020 Apr 29. PMID 32423584
- [Result] Spinner CD, Gottlieb RL, Criner GJ, Arribas Lopez JR, Cattelan AM, Soriano Viladomiu A, Ogbuagu O, Malhotra P, Mullane KM, Castagna A, Chai LYA, Roestenberg M, Tsang OTY, Bernasconi E, Le Turnier P, Chang SC, SenGupta D, Hyland RH, Osinusi AO, Cao H, Blair C, Wang H, Gaggar A, Brainard DM, McPhail MJ, Bhagani S, Ahn MY, Sanyal AJ, Huhn G, Marty FM; GS-US-540-5774 Investigators. Effect of Remdesivir vs Standard Care on Clinical Status at 11 Days in Patients With Moderate COVID-19: A Randomized Clinical Trial. JAMA. 2020 Sep 15;324(11):1048-1057. doi: 10.1001/jama.2020.16349. PMID 32821939
- [Result] Garibaldi BT, Wang K, Robinson ML, Zeger SL, Bandeen-Roche K, Wang MC, Alexander GC, Gupta A, Bollinger R, Xu Y. Comparison of Time to Clinical Improvement With vs Without Remdesivir Treatment in Hospitalized Patients With COVID-19. JAMA Netw Open. 2021 Mar 1;4(3):e213071. doi: 10.1001/jamanetworkopen.2021.3071. PMID 33760094
- [Result] Ortolan A, Lorenzin M, Felicetti M, Doria A, Ramonda R. Does gender influence clinical expression and disease outcomes in COVID-19? A systematic review and meta-analysis. Int J Infect Dis. 2020 Oct;99:496-504. doi: 10.1016/j.ijid.2020.07.076. Epub 2020 Aug 12. PMID 32800858
- [Result] Matthay MA, Thompson BT. Dexamethasone in hospitalised patients with COVID-19: addressing uncertainties. Lancet Respir Med. 2020 Dec;8(12):1170-1172. doi: 10.1016/S2213-2600(20)30503-8. Epub 2020 Oct 29. No abstract available. PMID 33129421
- [Result] Gregory JM, Slaughter JC, Duffus SH, Smith TJ, LeStourgeon LM, Jaser SS, McCoy AB, Luther JM, Giovannetti ER, Boeder S, Pettus JH, Moore DJ. COVID-19 Severity Is Tripled in the Diabetes Community: A Prospective Analysis of the Pandemic's Impact in Type 1 and Type 2 Diabetes. Diabetes Care. 2021 Feb;44(2):526-532. doi: 10.2337/dc20-2260. Epub 2020 Dec 2. PMID 33268335
- [Result] Wang S, Ma P, Zhang S, Song S, Wang Z, Ma Y, Xu J, Wu F, Duan L, Yin Z, Luo H, Xiong N, Xu M, Zeng T, Jin Y. Fasting blood glucose at admission is an independent predictor for 28-day mortality in patients with COVID-19 without previous diagnosis of diabetes: a multi-centre retrospective study. Diabetologia. 2020 Oct;63(10):2102-2111. doi: 10.1007/s00125-020-05209-1. Epub 2020 Jul 10. PMID 32647915
- [Result] Singh AK, Singh R, Joshi SR, Misra A. Mucormycosis in COVID-19: A systematic review of cases reported worldwide and in India. Diabetes Metab Syndr. 2021 Jul-Aug;15(4):102146. doi: 10.1016/j.dsx.2021.05.019. Epub 2021 May 21. PMID 34192610
- [Result] WHO Solidarity Trial Consortium; Pan H, Peto R, Henao-Restrepo AM, Preziosi MP, Sathiyamoorthy V, Abdool Karim Q, Alejandria MM, Hernandez Garcia C, Kieny MP, Malekzadeh R, Murthy S, Reddy KS, Roses Periago M, Abi Hanna P, Ader F, Al-Bader AM, Alhasawi A, Allum E, Alotaibi A, Alvarez-Moreno CA, Appadoo S, Asiri A, Aukrust P, Barratt-Due A, Bellani S, Branca M, Cappel-Porter HBC, Cerrato N, Chow TS, Como N, Eustace J, Garcia PJ, Godbole S, Gotuzzo E, Griskevicius L, Hamra R, Hassan M, Hassany M, Hutton D, Irmansyah I, Jancoriene L, Kirwan J, Kumar S, Lennon P, Lopardo G, Lydon P, Magrini N, Maguire T, Manevska S, Manuel O, McGinty S, Medina MT, Mesa Rubio ML, Miranda-Montoya MC, Nel J, Nunes EP, Perola M, Portoles A, Rasmin MR, Raza A, Rees H, Reges PPS, Rogers CA, Salami K, Salvadori MI, Sinani N, Sterne JAC, Stevanovikj M, Tacconelli E, Tikkinen KAO, Trelle S, Zaid H, Rottingen JA, Swaminathan S. Repurposed Antiviral Drugs for Covid-19 - Interim WHO Solidarity Trial Results. N Engl J Med. 2021 Feb 11;384(6):497-511. doi: 10.1056/NEJMoa2023184. Epub 2020 Dec 2. PMID 33264556
- [Result] Wijaya I, Andhika R, Huang I, Purwiga A, Budiman KY, Bashari MH, Reniarti L, Roesli RMA. The use of Janus Kinase inhibitors in hospitalized patients with COVID-19: Systematic review and meta-analysis. Clin Epidemiol Glob Health. 2021 Jul-Sep;11:100755. doi: 10.1016/j.cegh.2021.100755. Epub 2021 May 2. PMID 33969237
- [Result] Chen CX, Wang JJ, Li H, Yuan LT, Gale RP, Liang Y. JAK-inhibitors for coronavirus disease-2019 (COVID-19): a meta-analysis. Leukemia. 2021 Sep;35(9):2616-2620. doi: 10.1038/s41375-021-01266-6. Epub 2021 May 14. PMID 33990684
- [Result] Guimaraes PO, Quirk D, Furtado RH, Maia LN, Saraiva JF, Antunes MO, Kalil Filho R, Junior VM, Soeiro AM, Tognon AP, Veiga VC, Martins PA, Moia DDF, Sampaio BS, Assis SRL, Soares RVP, Piano LPA, Castilho K, Momesso RGRAP, Monfardini F, Guimaraes HP, Ponce de Leon D, Dulcine M, Pinheiro MRT, Gunay LM, Deuring JJ, Rizzo LV, Koncz T, Berwanger O; STOP-COVID Trial Investigators. Tofacitinib in Patients Hospitalized with Covid-19 Pneumonia. N Engl J Med. 2021 Jul 29;385(5):406-415. doi: 10.1056/NEJMoa2101643. Epub 2021 Jun 16. PMID 34133856